CLINICAL TRIAL: NCT03534167
Title: Mobile Phone and Internet-Based Intervention for Vulnerable Youth
Brief Title: TODAY! A Mobile App Study
Acronym: TODAY!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Diane Chen, Medical Psychologist, Division of Adolescent Medicine, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-1540
Record Dates: First submitted 2018-05-04; First posted 2018-05-23 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Depression, Anxiety
Keywords: depression; anxiety; gay; youth; Cognitive Behavior Therapy
MeSH Terms: conditions — Depression; Anxiety Disorders; Homosexuality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TODAY! App and Coaching (Experimental): RCT participants will be randomized into a 10-week intervention condition during which they will receive the CBT modules through the TODAY! app. In addition to the mobile app, participants will receive coaching from the study Coach who is trained in Motivational Interviewing principles. Participants will complete mood and behavior assessments at 4 time-points over the course of 22 weeks.
  Interventions: Behavioral: TODAY! App and Coaching
- Referrals (No Intervention): RCT participants will be randomized into a 10-week wait-list control condition and will be provided with and encouraged to use mental health and lesbian, gay, bisexual, queer (LGBQ) referrals and resources in the community. Participants will complete mood and behavior assessments at 4 time-points over the course of 22 weeks. After the 22-week post intervention follow-up, control group participants will have the option to receive the intervention, however they will not be administered follow-up assessments or given coaching.

INTERVENTIONS:
Behavioral: TODAY! App and Coaching — The TODAY! app uses the skill building structure of Cognitive Behavior Therapy (CBT). The intervention will be divided into "modules," each devoted to a particular skill. Skills addressed within the intervention include increasing social support, engaging in goal-driven behaviors and reducing mood-driven (i.e., avoidance) behaviors, seeking out positive activities, replacing cognitive distortions with more adaptive thinking styles, improving problem-solving skills, reducing avoidance patterns, and increasing alternate coping strategies. The intervention will be supplemented with brief human contact in the form of a motivational coach. The Coach will be trained on the Motivational Interviewing principles upon which the coaching protocol is based.
  Arms: TODAY! App and Coaching

SUMMARY:
The aim of this study is to conduct a small randomized controlled trial (RCT) for a 10-week mobile phone intervention using principles of Cognitive Behavior Therapy to target general and minority stressors and treat anxiety and depression in young men romantically/sexually attracted to men.

DETAILED DESCRIPTION:
Investigators will conduct a double-arm RCT to develop the infrastructure and collection of data needed to power a larger RCT (e.g., rates of consent, retention rates). Clinical outcomes will be assessed for the purpose of detecting unexpected deterioration. Investigators will also collect usability feedback regarding the intervention which may be used to refine the treatment. Usage data will be used to identify under-used lessons and tools and improve their usefulness/appeal. Compliance with assessments will be monitored and used to improve retention protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Were assigned male at birth and identify as a man
2. Report romantic/sexual attraction to men;
3. Ages 14-24 years;
4. Resides in the Chicago metro area (i.e., Chicago or suburbs of Cook County)
5. Presents with clinically significant depressive or anxiety symptoms, per a 10+ on the PHQ-9 or 5+ on the GAD-7
6. Currently owns a mobile phone that is compatible with the intervention application, and believes they will be able to keep using this mobile phone for the next 10 weeks
7. Fluent in English.

Exclusion Criteria:

1. Has visual, hearing, voice, or motor impairment that would prevent completion of study procedures or use of the Internet or mobile phone.
2. Per self-reported history or the Mini-International Neuropsychiatric Interview (MINI) 7 (Adult version for participants ages 17-24 years and Kid version for ages 14-16 years), has ever been diagnosed with a psychotic disorder or bipolar disorder, or is currently diagnosed with obsessive compulsive disorder, or has been diagnosed in the past two years with posttraumatic stress disorder, dissociative disorder, or eating disorder; or evidences another condition that indicates this intervention may be insufficient to meet the youth's needs. If substance abuse disorder is currently present, PI or designated individual will use clinical judgement to determine whether severity/impairment related to substance use indicates this intervention may be insufficient to meet the youth's needs.
3. Has been hospitalized for psychiatric reasons or has attempted suicide in the last year, or has a score of 4 or more (i.e., "high" to "severe" suicidality) on the Columbia Suicide Severity Rating Scale, or reports non-suicidal self-injury of a nature that suggests this intervention may be insufficient to meet the youth's needs.
4. Is concurrently participating in another behavioral intervention research study
5. Reports currently being in DCFS custody and under 21.
6. Reports currently being in psychotherapy.
7. Initiation, discontinuation, or adjustment of antidepressant medication in the past 4 weeks. Individuals excluded solely for this reason will be allowed to retake the baseline assessments (and be compensated accordingly) to determine eligibility after they have been on a stable antidepressant regimen for 4 weeks, if the study is still enrolling at that time.
8. Less than an 8th grade reading level.
9. Does not have an email address and does not obtain one within 1 week of the telephone screening.

Ages: 14 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Cisgender men (Assigned male at birth and identify as a man)
Enrollment: 22 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ) 9-items | Assessed at baseline, 5 weeks, 10 weeks and 22 weeks
  The PHQ-9 is a brief validated depression module. This study will measure change in PHQ-9 scores.
Change in Generalized Anxiety Disorder (GAD) 7-item Questionnaire | Assessed at baseline, 5 weeks, 10 weeks and 22 weeks
  The GAD-7 is a brief measure assessing anxiety. This study will measure change in GAD-7 scores.

SECONDARY OUTCOMES:
Usability feedback | Assessed at baseline, 5 weeks, 10 weeks and 22 weeks. Data regarding usage will be generated on the back end
  Usability feedback data will be qualitative, and it may be used to refine intervention components rather than formal analysis. Data entered by the participant into the mobile phone application may also be analyzed for utilization patterns and internal improvements.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Chen, Ph.D., Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Determination made by PI on a case by case basis